CLINICAL TRIAL: NCT05757882
Title: Comparison of Gastric Ultrasound for Reduction of Fasting Time in Children for Sedation
Brief Title: Reducing Fasting Time in Children for Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunah Cho, MD (Other)
Collaborators: Samsung Medical Center (Other)
Responsible Party: Sponsor-Investigator, Eunah Cho, MD, Assistant Professor, Kangbuk Samsung Hospital
Organization: Kangbuk Samsung Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NPO2
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4H (Active Comparator): Participants who are following the standard fasting time (4 hours).
  Interventions: Other: 4 hours of fasting time
- 2H (Experimental): Participants who are following minimized fasting time (2 hours)
  Interventions: Other: 2 hours of fasting time

INTERVENTIONS:
Other: 4 hours of fasting time — Oral intake is not allowed for 4 hours before sedation including water.
  Arms: 4H
Other: 2 hours of fasting time — Oral intake is not allowed for 2 hours before sedation including water.
  Arms: 2H

SUMMARY:
Patients are asked to be fasted for certain period of time before sedation to reduce the risk of pulmonary aspiration. However, fasting can be harmful, especially in children who has smaller reserves of energy and fluids compared to the adults. Prolonged fasting may increase nausea, vomiting, dehydration, and hypoglycemia. Therefore, it is important to minimize prolonged fasting time in pediatric patients.

This study is aimed to investigate the safety of minimal fasting time (2 hours) compared to the standard fasting time (4 hours) with gastric ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients aged under 36 months
* scheduled for elective cardiac echocardiography

Exclusion Criteria:

* patients with disease that delay gastric emptying
* patients taking medication that delay gastric emptying
* structural deformities, or abnormalities that interrupt gastric ultrasound
* refuse to participate in the study
* sedation is failed or impossible

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Risk of aspiration | 10 minutes before sedation
  Gastric antral cross-sectional area assessed with gastric ultrasound

SECONDARY OUTCOMES:
The incidence of complications | 10 minutes after sedation
  he incidence of major (pulmonary aspiration, aspiration pneumonia) and minor complications (nausea and vomiting, dehydration) between two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinyoung Song, Seoul, Gangnam, South Korea

IPD SHARING:
Plan to Share IPD: Undecided